CLINICAL TRIAL: NCT00892918
Title: A Randomized Clinical Trial Comparing the Effect of Moxifloxacin Versus Gatifloxacin Following Pterygium Excision on Corneal Epithelial Healing and Epithelial Toxicity.
Brief Title: Effect of Moxifloxacin Versus Gatifloxacin on Corneal Epithelium Following Pterygium Excision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator-Sponsor: Dr. Segev Fani, MD, Meir Medical Center, Kfar Saba, ISRAEL
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PVZ-001
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-03

CONDITIONS: Primary Pterygium
Keywords: pterygium; gatifloxacin; moxifloxacin; corneal epithelial defect
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Active Comparator): About 20 patients treated by Moxifloxacin ophthalmic solution 0.5% (Vigamox) 4 times a day (one drop each time) after pterygium excision with Mitomycin C application.
  Interventions: Drug: Moxifloxacin ophthalmic solution 0.5% ; Gatifloxacin ophthalmic solution 0.3%
- Gatifloxacin (Active Comparator): About 20 patients treated by Gatifloxacin ophthalmic solution 0.3% (Zymar) 4 times a day (one drop each time) after pterygium excision with Mitomycin C application.
  Interventions: Drug: Moxifloxacin ophthalmic solution 0.5% ; Gatifloxacin ophthalmic solution 0.3%

INTERVENTIONS:
Drug: Moxifloxacin ophthalmic solution 0.5% ; Gatifloxacin ophthalmic solution 0.3% — Each drug will be given 4 times a day, 1 drop each time to the operated eye, for 21 days.

SUMMARY:
The purpose of this study is to determine whether there is a difference in corneal epithelial healing rate and/or toxicity following pterygium excision, between eyes treated post-operatively by moxifloxacin(VIGAMOX)versus gatifloxacin (ZYMAR).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of primary pterygium with a clinical indication for surgery
2. informed consent

Exclusion Criteria:

1. known allergic reaction to fluoroquinolones.
2. secondary\recurrent pterygium or clinical suspected conjunctival tumor.
3. eye surgery in the last 6 months.
4. eye disorders: severe dry eye syndrome, ocular surface diseases, glaucoma, recurrent corneal erosions, chronic corneal diseases, after chemical burn.
5. low compliance.
6. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
rate of corneal epithelial defect closure | 21 days

SECONDARY OUTCOMES:
toxicity findings: punctate keratitis, inferior conjunctival hyperemia, conjunctival papillary reaction | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Fani Segev, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Cutarelli PE, Lass JH, Lazarus HM, Putman SC, Jacobs MR. Topical fluoroquinolones: antimicrobial activity and in vitro corneal epithelial toxicity. Curr Eye Res. 1991 Jun;10(6):557-63. doi: 10.3109/02713689109001764. PMID 1893771
- [Background] Kovoor TA, Kim AS, McCulley JP, Cavanagh HD, Jester JV, Bugde AC, Petroll WM. Evaluation of the corneal effects of topical ophthalmic fluoroquinolones using in vivo confocal microscopy. Eye Contact Lens. 2004 Apr;30(2):90-4. doi: 10.1097/01.icl.00000117255.97190.98. PMID 15260356
- [Background] Reviglio VE, Hakim MA, Song JK, O'Brien TP. Effect of topical fluoroquinolones on the expression of matrix metalloproteinases in the cornea. BMC Ophthalmol. 2003 Oct 6;3:10. doi: 10.1186/1471-2415-3-10. PMID 14529574
- [Background] Patel GM, Chuang AZ, Kiang E, Ramesh N, Mitra S, Yee RW. Epithelial healing rates with topical ciprofloxacin, ofloxacin, and ofloxacin with artificial tears after photorefractive keratectomy. J Cataract Refract Surg. 2000 May;26(5):690-4. doi: 10.1016/s0886-3350(00)00411-9. PMID 10831898
- [Background] Moreira LB, Lee RF, de Oliveira C, LaBree L, McDonnell PJ. Effect of topical fluoroquinolones on corneal re-epithelialization after excimer laser keratectomy. J Cataract Refract Surg. 1997 Jul-Aug;23(6):845-8. doi: 10.1016/s0886-3350(97)80241-6. PMID 9292666
- [Background] Burka JM, Bower KS, Vanroekel RC, Stutzman RD, Kuzmowych CP, Howard RS. The effect of fourth-generation fluoroquinolones gatifloxacin and moxifloxacin on epithelial healing following photorefractive keratectomy. Am J Ophthalmol. 2005 Jul;140(1):83-7. doi: 10.1016/j.ajo.2005.02.037. PMID 15953577
- [Background] Moshirfar M, Marx DP, Kumar R. The effect of the fourth-generation fluoroquinolones on corneal reepithelialization after penetrating keratoplasty. Cornea. 2005 Oct;24(7):833-6. doi: 10.1097/01.ico.0000157420.11448.d4. PMID 16160500
- [Background] Herrygers LA, Noecker RJ, Lane LC, Levine JM. Comparison of corneal surface effects of gatifloxacin and moxifloxacin using intensive and prolonged dosing protocols. Cornea. 2005 Jan;24(1):66-71. doi: 10.1097/01.ico.0000134182.09569.e1. PMID 15604869
- [Background] Barequet IS, Habot-Wilner Z, Lavinsky F, Ziv H, Belkin M, Rosner M. Effect of fourth-generation fluoroquinolones on the healing rate of corneal erosions in an animal model. Cornea. 2007 Jun;26(5):606-9. doi: 10.1097/ICO.0b013e318041f08e. PMID 17525660